CLINICAL TRIAL: NCT06871566
Title: Artificial Intelligence-Supported Occupational Therapy Program on Handwriting Skills in Children at Risk for Developmental Coordination Disorder: Randomized Controlled Trial
Brief Title: AI-Supported Occupational Therapy for Handwriting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güleser Güney Yılmaz, PhD Occupational Therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-242
Record Dates: First submitted 2025-01-22; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Occupational Therapy
Keywords: Artifical intellegence; occupational therapy; developmental coordination disorders; handwriting; rehabilitation
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children at Risk for Developmental Coordination Disorder
  Interventions: Other: Artificial Intelligence-Supported Occupational Therapy Program
- Control group (No Intervention): Children at Risk for Developmental Coordination Disorder

INTERVENTIONS:
Other: Artificial Intelligence-Supported Occupational Therapy Program — The AI-supported occupational therapy program was individually implemented by an occupational therapist over 8 weeks, with 2 sessions per week, each lasting 45 minutes. A touchscreen tablet, touch pen, and external camera were utilized during the sessions. At the beginning of the program, technological devices and artificial intelligence tools were introduced to the children. For the goals and detailed intervention program of the 8-week schedule
  Arms: Study group

SUMMARY:
Aim: This study investigates the impact of an AI-supported occupational therapy program, developed using the Model of Human Occupation (MOHO), on handwriting skills in children at risk for Developmental Coordination Disorder (DCD).

Method: A randomized controlled trial was conducted with 42 children aged 8-12 years, identified as being at risk for DCD using the Developmental Coordination Disorder Questionnaire (DCDQ). Participants were randomized into an intervention group (n=21) and a control group (n=21). The intervention group received an AI-supported occupational therapy program twice weekly for 8 weeks. Handwriting performance was assessed pre- and post-intervention using the Minnesota Handwriting Assessment (MHA).

Keywords: artificial intelligence, occupational

ELIGIBILITY:
Inclusion Criteria:

1. being between the ages of 8-12 years
2. being at risk for DCD according to the Developmental Coordination Disorder Questionnaire (DCDQ)
3. having the ability to understand the questionnaires
4. continuing formal education
5. having similar motor skill performance (having similar results from the Bruininks-Oseretsky Motor Proficiency Test 2 Brief Form (BOT2-BF)) and having similar visual perception level (having similar results from the Motor-Free Visual Perception Test-3(MVPT-3)

Exclusion Criteria:

(1) having another neurodevelopmental, orthopedic and chronic problem (2) continuing any rehabilitation program

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Minnesota Handwriting Assessment | Two assessments, one week before the intervention and one week after the intervention was completed
  (MHA) assesses six categories of handwriting, including legibility, form, alignment, size, spacing and writing speed. The MHA consists of words that include all letters of the Turkish alphabet at least once and consist of 34 letters in total, and can be understood by children at the primary school level 23. In the test application, children copy this word sequence written on the paper to the marked line immediately below. In the scoring phase, the length of 1/16 inch (0.15 cm) is taken as a basis and all deviations, proportions between letters and within letters are evaluated by measuring this length with a ruler. The lowest score in each category of the MHA is 0 and the highest score is 34 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Güleser Güney Yılmaz, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
This study investigates the impact of an AI-supported occupational therapy program, developed using the Model of Human Occupation (MOHO), on handwriting skills in children at risk for Developmental Coordination Disorder (DCD).